CLINICAL TRIAL: NCT06320002
Title: Improving Biopsychosocial Outcomes With a Communication Intervention for Patients Undergoing Fecal Ostomy Surgery
Brief Title: Communication Intervention for Fecal Ostomy Surgery
Acronym: CI-oSurg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christy E. Cauley, MD, MPH, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023P003564
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Surgery; Colostomy Stoma; Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal ostomy surgery participants receiving the CI-oSurg (Experimental): This arm will include patients who are undergoing or have undergone fecal ostomy surgery and surgical clinicians caring for the patients who will receive the CI-oSurg intervention.
  Interventions: Behavioral: Communication Intervention for fecal ostomy surgery

INTERVENTIONS:
Behavioral: Communication Intervention for fecal ostomy surgery — This is a educational video-based supportive intervention to address practical skills and adaptation to life with a fecal ostomy

SUMMARY:
In this study the investigators will evaluate the acceptability of a communication intervention for fecal ostomy surgery (CI-oSurg) to address the needs of adults who are undergoing fecal ostomy surgery. The investigators will recruit 24 patients and 4 clinicians (surgical nurses, wound ostomy nurses). At least half of patients are 65 years or older to understand the unique needs of older adults recovering from fecal ostomy surgery that might impact intervention acceptability. Questionnaires will be administered at two time-points for patient participants: upon study start and 4 weeks after exposure to the intervention.

DETAILED DESCRIPTION:
In this study the investigators are trying to understand the feasibility and acceptability of a psychologically informed communication guide for fecal ostomy Surgery with the overall goal of improving biopsychosocial outcomes of patients undergoing fecal ostomy surgery.

An estimated 100,000 people in the US undergo fecal ostomy surgery (colostomy or ileostomy) each year, frequently to address severe symptoms (i.e., obstruction, perforation, and incontinence) due to colorectal cancer, diverticulitis, and pelvic floor dysfunction. Complication rates after fecal ostomy surgery are high (up to 37%) with negative effects on patient and family quality of life. Surgeons do not traditionally identify and address health outcomes patients with serious illness prioritize when making treatment decisions, such as caregiver burden, loss of independence and psychosocial function. Communicating this information is key to address patient anxiety when facing major surgery and ensure caregiver preparedness among patients and families considering fecal ostomy surgery.

Current surgical guidelines support the use of preoperative communication and education interventions to improve psychosocial adjustment after fecal ostomy surgery based on expert opinion. However, little evidence exists evaluating the impact of communication interventions or content needs of patients undergoing fecal ostomy surgery or their family. Despite these guidelines, a recent study notes that inadequate ostomy education remains a frequent concern among patients undergoing fecal ostomy surgery. Furthermore, patients' perception of inadequate education is associated with poor emotional, social, and marital outcomes after surgery. There is a critical need to address this deficit in communication quality between patients undergoing fecal ostomy surgery, their family, and surgical care providers. Our guiding hypothesis is that development of a Communication Intervention for fecal ostomy Surgery (CI-oSurg) is acceptable to patients and clinicians, and will ultimately reduce patient distress and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. English fluency and literacy
3. Patient planned to undergo elective fecal ostomy surgery

Exclusion Criteria:

1. Deemed inappropriate by the surgery team
2. Unable to provide consent due to severe cognitive impairment or physiologic status (septic shock/intubated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability | 4 weeks after the intervention
  The intervention acceptability will be assessed by cognitive interviews with participants

SECONDARY OUTCOMES:
Intervention Usability | 4 weeks after intervention use
  The intervention usability will be assessed by cognitive interviews with participants

OTHER OUTCOMES:
Emotional Distress | baseline and 4 weeks after intervention
  Exploratory outcome of Distress reported by patients from 0-10
World Health Organization Brief quality of life evaluation | baseline and 4 weeks after intervention
  There are 26 questions with scores ranging from 1-5. For 23 questions higher score is better and for 3 questions a lower score is better.
Hospital Anxiety and Depression Scale | baseline and 4 weeks after intervention
  This survey has 14 questions with scores ranging from 1-4. A higher score is better.
Therapy Evaluation Form | baseline and 4 weeks after intervention
  This survey has 6 questions with scores ranging from 1-9. A higher score is better.
Client Satisfaction Questionnaire | baseline and 4 weeks after intervention
  This survey has 8 questions with scores ranging from 1-4. A higher score is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data of qualitative interviews will be shared with other researchers upon request.

REFERENCES:
- [Derived] Cauley CE, Rubio A, Brindle M, Cooper Z, Vranceanu AM, Ritchie CS. A Video-Based Communication Intervention for Fecal Ostomy Surgery (CI-oSurg): Protocol for Open Pilot Testing to Improve Intervention Acceptability and Feasibility. JMIR Res Protoc. 2024 Nov 15;13:e60575. doi: 10.2196/60575. PMID 39546348